CLINICAL TRIAL: NCT01880515
Title: Phase II, Open-label, Single Blind, Randomised Clinical Trial With Tetracycline as a Prophylaxis for Rash and Dermatological Recommendations Versus Dermatological Recommendations in Patients With NSCLC Receiving Treatment With BIBW 2992
Brief Title: Tetracycline as a Prophylaxis for Rash in Patients With NSCLC Receiving Treatment With BIBW2992 (Afatinib)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Oscar Gerardo Arrieta Rodríguez, M.D., M.Sc., Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TEPR-BIBW2992
Record Dates: First submitted 2013-05-31; First posted 2013-06-19 (Estimated); Results first posted 2017-04-12 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-04

CONDITIONS: Skin Rash; Lung Cancer
Keywords: Lung cancer; BIBW 2992; Skin Rash; Tetracycline; Afatinib
MeSH Terms: conditions — Exanthema; Lung Neoplasms | interventions — Tetracycline

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetracycline (Experimental): Patients will receive tetracycline 250mg every 12 hours for 1 month plus general dermatological recommendations (sunscreen and emollient cream)
  Interventions: Drug: Tetracycline
- No Tetracycline (No Intervention): This arm only with general dermatologic recommendations. Patients in this arm can receive tetracycline after week 4 of assessment only if rash grade 3-4 occur

INTERVENTIONS:
Drug: Tetracycline — The experimental group will receive tetracycline 250mg every 12 hours for 1 month the same day at initiation of BIBW2992 whereas the non-intervention group will recieve general dermatological recomendations while on treatment with BIBW2992.
  Other Names: Tetracycline hydrocloride; Tetrex®
  Arms: Tetracycline

SUMMARY:
1. Advanced NSCLC has a poor prognosis and the positive impact of chemotherapy is limited by the development of intrinsic and acquired resistance.
2. Over the past decade, less toxic agents such as the innovative targeted therapies, i.e. erlotinib or gefitinib, have the potential to improve the effectiveness and keep a good quality of life with a low toxicity
3. BIBW2992 (afatinib), an aniline-quinazoline, is an epidermal growth factor receptor (EGFR) and human epidermal growth factor receptor 2 (HER-2) irreversible inhibitor, and it has activity against erlotinib-resistant isoforms having mutations in EGFR and HER-2.
4. This molecule has shown benefits as a single agent in pre-treated patients who have progressed despite platinum-based chemotherapy, with a minimal toxicity compared to chemotherapy.
5. BIBW2992 is associated with adverse effects similar to those for erlotinib and gefitinib, such as rash and diarrhea. These symptoms can reduce the quality of life (QL) in patients and lead to inconsistent EGFR inhibitor dose administration
6. There is not a standard treatment for rash. However, case reports have tried to demonstrate the benefit in the treatment of these cutaneous injuries obtained with alcohol-free emollients, sunscreen with titanium dioxide or antibiotic (topic or oral) treatment regimens that include clindamycin or doxycycline, as well as anti-inflammatory drugs such as steroids and isotretinoin.
7. In order to reduce the incidence and severity of cutaneous toxicities, we will compare the prophylactic antibiotic treatment using tetracycline and general dermatological recommendations versus using only dermatological recommendations, in patients initiating the treatment with BIBW2992.

DETAILED DESCRIPTION:
Case reports have tried to demonstrate the benefit in the treatment of rash obtained with: alcohol-free emollients used 2-3 times daily, sunscreen with titanium dioxide or zinc oxide with a skin protection factor (SPF) greater than 15, topic or oral antibiotic regimens (such as clindamycin, metronidazole, tetracyclines) when there is secondary infection as well as steroidal anti-inflammatory drugs (betamethasone, triamcinolone) and isotretinoin.

The objective of this project is to evaluate whether the prophylactic treatment with tetracycline can reduce dermatological toxicities such as rash, induced by the EGFR and HER-2 tyrosine kinase inhibitor BIBW 2992 in patients with non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of non-operable, locally advanced, recurrent or metastatic, histologically or cytologically documented non-small cell lung cancer (stage IIIB or IV).

  * Patients should have an evidence of measurable disease.
  * 18 years or older
  * Eastern Cooperative Oncology Group - Performance Status 0-3
  * At least 12 weeks of life expectancy
  * Patients with non-small cell lung cancer stages IIIB/IV who have received at least one cycle of platinum-based, first or second line systemic standard chemotherapy, and have a documented failure for this treatment.
  * More than 2 previous chemotherapy regimens are not allowed. The patients should have recovered from any toxic effect and at least 2 weeks should have elapsed from last dose before their entry (14 days for vinorelbine and other vinca alkaloids or gemcitabine). Patients who in the investigator's opinion are fully recovered from surgery for at least 4 weeks may also be considered for the study. Patients should have recovered from any severe toxicity (CTC > 1) caused by any previous therapy.
  * Granulocyte count > 1.5x 109/L and platelet count > 100x 109/L.
  * Serum bilirubin > 1.5 upper limit of normal (ULN)
  * AST and/or ALT > 2 ULN (or >5 x ULN when clearly attributable to presence of hepatic metastases).
  * Serum creatinine > 1.5 ULN or creatinine clearance < 60 mL/min
  * Capability to fulfill the study and follow-up procedures.
  * A negative pregnancy test should be obtained from all women of childbearing potential within 72 hours previous to therapy beginning.
  * Patients of reproductive potential should use effective contraceptive methods.
  * Written (signed) informed consent to participate in the study

Exclusion Criteria:

* Patients allergic to the antibiotic therapy used.
* Any unsteady systemic disease (including active infection, uncontrolled hypertension, unsteady angina, congestive cardiac failure, hepatic, renal or metabolic disease).
* A previous treatment using a systemic anti-tumor therapy with EGFR inhibitors (tyrosine kinase inhibitors).
* Any other malignant pathology within 5 previous years (except for carcinoma in situ of cervix or basal-cell type skin cancer appropriately treated).
* Patients with cerebral metastases or spinal marrow compression recently diagnosed and/or definitely surgery and/or radiation naïve-treatment patients are excluded. Those with previously diagnosed and treated metastasis to Central Nervous System (CNS) or spinal marrow compression, having an evidence of steady disease (clinically steady in imaging studies) are accepted for at least 2 months.
* Any significant ophthalmologic abnormality, especially severe dry-eye syndrome, keratoconjunctivitis sicca, Sjögren's syndrome, severe exposure keratitis and any other disorder that may increase the risk for corneal epithelial injure. Contact lens use during the study is not recommended. The decision to continue to use contact lens should be discussed with the oncologist responsible for patient treatment and the ophthalmologist.
* Patients who cannot take oral medication, requiring intravenous nutrition, who underwent previous surgical procedures affecting absorption, or with active peptic ulcer.
* Nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Arrieta, M.D., M.Sc., Principal Investigator — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico

REFERENCES:
- [Background] Modjtahedi H, Dean C. The receptor for EGF and its ligands - expression, prognostic value and target for therapy in cancer (review). Int J Oncol. 1994 Feb;4(2):277-96. doi: 10.3892/ijo.4.2.277. PMID 21566922
- [Background] Salomon DS, Brandt R, Ciardiello F, Normanno N. Epidermal growth factor-related peptides and their receptors in human malignancies. Crit Rev Oncol Hematol. 1995 Jul;19(3):183-232. doi: 10.1016/1040-8428(94)00144-i. No abstract available. PMID 7612182
- [Background] Rusch V, Mendelsohn J, Dmitrovsky E. The epidermal growth factor receptor and its ligands as therapeutic targets in human tumors. Cytokine Growth Factor Rev. 1996 Aug;7(2):133-41. doi: 10.1016/1359-6101(96)00016-0. PMID 8899291
- [Background] Davies DE, Chamberlin SG. Targeting the epidermal growth factor receptor for therapy of carcinomas. Biochem Pharmacol. 1996 May 3;51(9):1101-10. doi: 10.1016/0006-2952(95)02232-5. PMID 8645330
- [Background] Eskens FA, Mom CH, Planting AS, Gietema JA, Amelsberg A, Huisman H, van Doorn L, Burger H, Stopfer P, Verweij J, de Vries EG. A phase I dose escalation study of BIBW 2992, an irreversible dual inhibitor of epidermal growth factor receptor 1 (EGFR) and 2 (HER2) tyrosine kinase in a 2-week on, 2-week off schedule in patients with advanced solid tumours. Br J Cancer. 2008 Jan 15;98(1):80-5. doi: 10.1038/sj.bjc.6604108. Epub 2007 Nov 20. PMID 18026190
- [Background] C. Yang, J. Shih, W. Su, Et.Al. A phase II study of BIBW 2992 in patients with adenocarcinoma of the lung and activating EGFR mutations (LUX-Lung 2).- J Clin Oncol 28: 15s, 2010 (Suppl; Abstr 7521).
- [Background] Yap TA, Vidal L, Adam J, Stephens P, Spicer J, Shaw H, Ang J, Temple G, Bell S, Shahidi M, Uttenreuther-Fischer M, Stopfer P, Futreal A, Calvert H, de Bono JS, Plummer R. Phase I trial of the irreversible EGFR and HER2 kinase inhibitor BIBW 2992 in patients with advanced solid tumors. J Clin Oncol. 2010 Sep 1;28(25):3965-72. doi: 10.1200/JCO.2009.26.7278. Epub 2010 Aug 2. PMID 20679611
- [Background] C. Yang, J. Shih, T. Chao, C. Tsai, Et.Al. Use of BIBW 2992, a novel irreversible EGFR/HER2 TKI, to induce regression in patients with adenocarcinoma of the lung and activating EGFR mutations: Preliminary results of a single-arm phase II clinical trial. J Clin Oncol 26: 2008
- [Background] Veale D, Ashcroft T, Marsh C, Gibson GJ, Harris AL. Epidermal growth factor receptors in non-small cell lung cancer. Br J Cancer. 1987 May;55(5):513-6. doi: 10.1038/bjc.1987.104. PMID 3038157
- [Background] Gatzemeier U, Pluzanska A, Szczesna A, Kaukel E, Roubec, Brennscheidt U, De Rosa F, Mueller B, Von Pawel J: Results of a phase III trial of erlotinib (OSI-774) combined with cisplatin and gemcitabine (GC) chemotherapy in advanced non-small cell lung cancer (NSCLC) ASCO Annual Meeting 2004 abstract number 7010
- [Background] Herbst RS, Prager D, Hermann R, Fehrenbacher L, Johnson BE, Sandler A, Kris MG, Tran HT, Klein P, Li X, Ramies D, Johnson DH, Miller VA; TRIBUTE Investigator Group. TRIBUTE: a phase III trial of erlotinib hydrochloride (OSI-774) combined with carboplatin and paclitaxel chemotherapy in advanced non-small-cell lung cancer. J Clin Oncol. 2005 Sep 1;23(25):5892-9. doi: 10.1200/JCO.2005.02.840. Epub 2005 Jul 25. PMID 16043829
- [Background] Li D, Ambrogio L, Shimamura T, Kubo S, Takahashi M, Chirieac LR, Padera RF, Shapiro GI, Baum A, Himmelsbach F, Rettig WJ, Meyerson M, Solca F, Greulich H, Wong KK. BIBW2992, an irreversible EGFR/HER2 inhibitor highly effective in preclinical lung cancer models. Oncogene. 2008 Aug 7;27(34):4702-11. doi: 10.1038/onc.2008.109. Epub 2008 Apr 14. PMID 18408761
- [Background] Sharma SV, Bell DW, Settleman J, Haber DA. Epidermal growth factor receptor mutations in lung cancer. Nat Rev Cancer. 2007 Mar;7(3):169-81. doi: 10.1038/nrc2088. PMID 17318210
- [Background] Kobayashi S, Boggon TJ, Dayaram T, Janne PA, Kocher O, Meyerson M, Johnson BE, Eck MJ, Tenen DG, Halmos B. EGFR mutation and resistance of non-small-cell lung cancer to gefitinib. N Engl J Med. 2005 Feb 24;352(8):786-92. doi: 10.1056/NEJMoa044238. PMID 15728811
- [Background] Maheswaran S, Sequist LV, Nagrath S, Ulkus L, Brannigan B, Collura CV, Inserra E, Diederichs S, Iafrate AJ, Bell DW, Digumarthy S, Muzikansky A, Irimia D, Settleman J, Tompkins RG, Lynch TJ, Toner M, Haber DA. Detection of mutations in EGFR in circulating lung-cancer cells. N Engl J Med. 2008 Jul 24;359(4):366-77. doi: 10.1056/NEJMoa0800668. Epub 2008 Jul 2. PMID 18596266
- [Background] Takezawa K, Okamoto I, Tanizaki J, Kuwata K, Yamaguchi H, Fukuoka M, Nishio K, Nakagawa K. Enhanced anticancer effect of the combination of BIBW2992 and thymidylate synthase-targeted agents in non-small cell lung cancer with the T790M mutation of epidermal growth factor receptor. Mol Cancer Ther. 2010 Jun;9(6):1647-56. doi: 10.1158/1535-7163.MCT-09-1009. Epub 2010 Jun 8. PMID 20530710
- [Background] Rudin CM, Liu W, Desai A, Karrison T, Jiang X, Janisch L, Das S, Ramirez J, Poonkuzhali B, Schuetz E, Fackenthal DL, Chen P, Armstrong DK, Brahmer JR, Fleming GF, Vokes EE, Carducci MA, Ratain MJ. Pharmacogenomic and pharmacokinetic determinants of erlotinib toxicity. J Clin Oncol. 2008 Mar 1;26(7):1119-27. doi: 10.1200/JCO.2007.13.1128. PMID 18309947
- [Background] Collen G., Vos L.E., Laurijsen A., Clasificación y tratamiento de los efectos secundarios de los inhibidorres del receptor de factor de crecimiento epidérmico (EGFR) en piel, pelo, uñas y mucosas. European Journal of Cancer. 2007, Vol 43: 845-851
- [Background] Lacouture ME. Mechanisms of cutaneous toxicities to EGFR inhibitors. Nat Rev Cancer. 2006 Oct;6(10):803-12. doi: 10.1038/nrc1970. PMID 16990857
- [Background] Topham E. Cutaneous manifestations of cancer and chemotherapy. Clin Med (Lond). 2009 Aug;9(4):375-9. doi: 10.7861/clinmedicine.9-4-375. No abstract available. PMID 19728518
- [Background] Wacker B, Nagrani T, Weinberg J, Witt K, Clark G, Cagnoni PJ. Correlation between development of rash and efficacy in patients treated with the epidermal growth factor receptor tyrosine kinase inhibitor erlotinib in two large phase III studies. Clin Cancer Res. 2007 Jul 1;13(13):3913-21. doi: 10.1158/1078-0432.CCR-06-2610. PMID 17606725
- [Background] Hammond-Thelin LA. Cutaneous reactions related to systemic immunomodulators and targeted therapeutics. Dermatol Clin. 2008 Jan;26(1):121-59, ix. doi: 10.1016/j.det.2007.08.010. PMID 18023775
- [Background] Hu JC, Sadeghi P, Pinter-Brown LC, Yashar S, Chiu MW. Cutaneous side effects of epidermal growth factor receptor inhibitors: clinical presentation, pathogenesis, and management. J Am Acad Dermatol. 2007 Feb;56(2):317-26. doi: 10.1016/j.jaad.2006.09.005. Epub 2006 Dec 1. PMID 17141360
- [Derived] Arrieta O, Vega-Gonzalez MT, Lopez-Macias D, Martinez-Hernandez JN, Bacon-Fonseca L, Macedo-Perez EO, Ramirez-Tirado LA, Flores-Estrada D, de la Garza-Salazar J. Randomized, open-label trial evaluating the preventive effect of tetracycline on afatinib induced-skin toxicities in non-small cell lung cancer patients. Lung Cancer. 2015 Jun;88(3):282-8. doi: 10.1016/j.lungcan.2015.03.019. Epub 2015 Mar 28. PMID 25882778

RESULTS

PARTICIPANT FLOW:
Groups:
- Tetracycline: Patients will receive tetracycline 250mg every 12 hours for 1 month plus general dermatological recommendations (sunscreen and emollient cream)
  Tetracycline: The experimental group will receive tetracycline 250mg every 12 hours for 1 month the same day at initiation of BIBW2992 (afatinib)
Period: Overall Study
Arm/Group | Tetracycline | No Tetracycline
Started | 53 | 54
Completed | 45 | 45
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 3 | 2
Not completed — Disease Progression | 5 | 7

BASELINE CHARACTERISTICS:
Population: A total of 107 patients were enrolled. Due to progression and lost to follow-up, only 90 patients were evaluated for dermatological toxicities. Forty five patients were assigned to receive reactive treatment; the other 45 received pre-emptive tetracycline.
Groups:
- Tetracycline: Patients will receive tetracycline 250mg every 12 hours for 1 month plus general dermatological recommendations
  Tetracycline: The experimental group will receive tetracycline 250mg every 12 hours for 1 month the same day at initiation of BIBW 2992
- Total: Total of all reporting groups
Arm/Group | Tetracycline | No Tetracycline | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (14) | 56.6 (14) | 57.05 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 66
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Mexico | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Participants Who Experienced Any Grade of Rash As Characterized By The Common Toxicity Criteria for Adverse Effects (CTCAE) V4.0
Description: Sum of participants who experienced any grade rash according to the Common Toxicity Criteria for Adverse Effects (CTCAE) V4.0, from the initiation of BIBW2992 compared to week 8.
Time Frame: Percentage of adverse events at week 8
Population: Forty five patients were assigned to receive reactive treatment; the other 45 received pre-emptive tetracycline.There were no differences among demographics, disease stage and dermatological baseline characteristics between treatment groups.
Measure: Number; unit: Percentage of Patients w/any grade rash
Groups:
- Tetracycline: Patients will receive tetracycline 250mg every 12 hours for 1 month plus general dermatological recommendations (sunscreen and emollient cream)
  Tetracycline: The experimental group will receive tetracycline 250mg every 12 hours for 1 month the same day at initiation of BIBW 2992
Arm/Group | Tetracycline | No Tetracycline
Number analyzed (Participants) | 45 | 45
Percentage of Patients w/any grade rash | 44.5 | 75.5
Statistical Analysis 1: Comparison: Tetracycline vs No Tetracycline; Test type: Superiority or Other; Risk Ratio (RR) = .4, 95% CI 2-sided [0.17 to 0.99]

2. Secondary Outcome: Quality of Life (QoL)
Description: A QoL questionnaire from European Organization for Research and Treatment of Cancer (EORTC) organization (Spanish version) will be performed at initiation of BIBW 2992 and then every month of follow-up until progression
Time Frame: from baseline to 6 months
Reporting Status: Not Posted, anticipated posting 2025-12

3. Secondary Outcome: Progression Free-survival
Description: The measure will be from the start of consumption to the first documented evidence of progression according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, or if patients still survive the measure will be made after 24 weeks
Time Frame: 24 weeks from baseline
Reporting Status: Not Posted, anticipated posting 2025-12

4. Secondary Outcome: Progression Free Survival
Description: From the start of consumption of BIBW 2992 to the date progression or last follow up
Time Frame: Participants will be followed for the duration of the treatment, an average of 8 weeks.
Population: We estimated the progression free survival with the Kaplan Meier method, and comparisons among groups were performed with the log-rank test.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tetracycline | No Tetracycline
Number analyzed (Participants) | 45 | 45
months | 8.1 [1.7 to 14.3] | 12.3 [7.1 to 17.5]
Statistical Analysis 1: Comparison: Tetracycline vs No Tetracycline; Test type: Superiority; p = 0.41, Log Rank

ADVERSE EVENTS:
Time Frame: All patients were followed-up, every two weeks for skin toxicities by a dermatologist since the start of treatment with afatinib, until the fourth week.
Arm/Group | Tetracycline | No Tetracycline
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No